CLINICAL TRIAL: NCT02126111
Title: Efficacy of a Depigmented Extract of Phleum in the Treatment of Local Allergic Rhinitis
Brief Title: Efficacy of a Depigmented Extract of Phleum in Local Allergic Rhinitis
Acronym: GRAMAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Plaza del Hospital Civil (Other)
Collaborators: Laboratorios Leti, S.L. (Industry)
Responsible Party: Principal Investigator, Miguel Blanca Gomez, Director Allergy Unit, Plaza del Hospital Civil
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MBG6043179
Record Dates: First submitted 2014-02-12; First posted 2014-04-29 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DEPIGOID phleum (Active Comparator): The active treatment arm receive active phleum pollen immunotherapy (Depigoid 100% phleum). Depigmented and polymerized allergen extract of Phleum pollen for subcutaneous injection.
  Interventions: Biological: DEPIGOID phleum
- DEPIGOID Placebo & DEPIGOID Phleum (Placebo Comparator): This arm receive DEPIGOID Placebo during the first year, and DEPIGOID Phleum during the second year of study.
  DEPIGOID Placebo contains the same composition as in the active DEPIGOID Phleum with the only difference being the exclusion of the phleum pollen allergen extract.
  Interventions: Biological: DEPIGOID phleum; Biological: DEPIGOID Placebo

INTERVENTIONS:
Biological: DEPIGOID phleum — Subcutaneous Immunotherapy with modified extract of Phleum pollen.
Biological: DEPIGOID Placebo — Placebo for subcutaneous administration
  Arms: DEPIGOID Placebo & DEPIGOID Phleum

SUMMARY:
The purpose of this study is evaluate the efficacy of a depigmented grass extract in the treatment of local allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Local allergic rhinitis with sensitization to grass pollen
* Skin prick test and serum specific IgE negative to grass pollen.
* Positive Nasal allergen provocation test (NAPT) to grass pollen and/or positive nasal specific IgE to grass pollen.
* Written informed consent

Exclusion Criteria:

* Immunological diseases
* Heart diseases that limit the use of adrenaline. For example, severe hypertension or treatment with beta-blockers.
* Treatment with beta-blockers
* Severe psychological disorders
* Severe atopic dermatitis
* FEV1 < 70% of reference value after treatment
* Hypersensitivity or intolerance to excipients and / or medication trial.
* Failure to adequately perform diagnostic tests or treatment.
* Sensitization to other allergens (perennial or seasonal) with clinical relevance for the subject and that may interfere in the evaluation of the response.
* Immunotherapy in the 5 years prior to their inclusion in the study.
* Pregnant women or at risk of pregnancy and lactating women.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2010-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Symptoms and medication scores comparison between active and placebo group | two years
  Patients were provided a diary to score the severity of their symptoms and the use of rescue medication during 4 weeks in two consecutive springs.
  Nasal symptoms of rhinorrhea, nasal congestion, sneezing, nasal itching, and ocular symptoms were recorded using a 4-point categorical scale from 0 to 3 (0: no symptoms, 1:mild, 2:moderate; 3:severe).
  The use of rescue medication was recorded in the patient diary according to the following score:
  Oral antihistamines (1 tablet = 1 point); intranasal corticosteroids (400mcg/day of beclometasone or equivalent = 1.4 points); and ocular antihistamines (1 dose = 1 point).

SECONDARY OUTCOMES:
Response to nasal allergen provocation test with phleum (NAPT-Phl) | two years
  The response to NAPT-Phl with increasing concentrations of phleum pratense (0.001-0.01-0.05-0.1 mcg/ml) will be evaluated by nasal symptoms and acoustic rhinometry.
Skin prick-test (SPT) with phleum. | 2 years
  Evaluation of SPT wheal size.
Intradermal test (IDT) with phleum | 2 years
  IDT wheal and erythema size.
FEV1 | 2 years
Quality of life questionnaire RQLQ | 2 years
Flow cytometry study for determination of IFN-gamma, IL-13, IL-5, IL-8, IL-10, IL-12, IL-2 in peripheral blood and nasal lavage | 2 years
Determination of tryptase, eosinophil cationic protein, IgG, IgG4, specific IgE to grass (Phl p1, Phl p5, Phl p7, Phl p12) in peripheral blood and nasal lavage. | 2 years
Heart rate | 2 years
Blood pressure | 2 years
Adverse events | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Blanca, MD, PhD, Principal Investigator — Hospital Regional Universitario, Málaga, Spain
Locations (2):
- Spain (2):
  - Hospital Infanta Leonor, Madrid, Madrid
  - Hospital Regional Universitario Carlos Haya, Málaga, Malaga

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rondon C, Blanca-Lopez N, Campo P, Mayorga C, Jurado-Escobar R, Torres MJ, Canto G, Blanca M. Specific immunotherapy in local allergic rhinitis: A randomized, double-blind placebo-controlled trial with Phleum pratense subcutaneous allergen immunotherapy. Allergy. 2018 Apr;73(4):905-915. doi: 10.1111/all.13350. Epub 2017 Nov 28. PMID 29168570